CLINICAL TRIAL: NCT04672850
Title: The Effect of Probiotic and Zinc Supplementation on the Common Cold in Healthy Adults
Brief Title: The Effect of Probiotic and Zinc Supplementation on the Common Cold
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lund University (Other)
Collaborators: Coradil AB (Unknown)
Responsible Party: Principal Investigator, Åsa Håkansson, Assoc. Prof., Lund University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Prozicold
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Rice flour
  Interventions: Dietary Supplement: Placebo
- Probiotic (Active Comparator): Probiotic bacteria, yeast, zinc and rice brand
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — The participants will consume 2 capsules daily for three months
  Arms: Probiotic
Dietary Supplement: Placebo — The participants will consume 2 capsules daily for three months
  Arms: Placebo

SUMMARY:
The purpose with this study is to investigate the preventative effect of a supplement containing a combination of probiotic bacteria and fungi as well as zinc on the common cold. The hypothesis is that it will shorten the duration, alleviate the severity of symptoms or even decrease the number of infectons during the intervention period. This study is a randomzed placebo controlled human study were healthy adults will consume the supplement for three months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Diagnosed gastrointestinal disorders
* Autoimmune diseases or immuno compromized
* Antibiotic treatment in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Symptoms severity | Three months
  Decrease in the severity of symptoms will be determined using a common cold questionnaire.

SECONDARY OUTCOMES:
Composition of gut and oral microbiome | Three months
  Change in gut and oral microbiome will be measured using 16SrRNA and 18SrRNA sequencing
IgA | Three months
  Changes in levels of IgA in saliva and/or feces will be measured using ELISA
Duration of symptoms | Three months
  Decrease in duration of cold will be determined using a common cold questionnaire
Number of colds | Three months
  Decrease in number of colds will be determined using a common cold questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Lunds universitet, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
Only group data will be shared